CLINICAL TRIAL: NCT07060001
Title: Evaluation of the Efficacy of Hypomethylating Agent Versus Standard Intensive Chemotherapy Induction Based on 5hmC - a Novel, Blood Epigenetic Marker for Assessing Measurable Residual Disease in Patients With Acute Myeloid Leukemia
Brief Title: Efficacy of Hypomethylating Agents vs. Intensive Chemotherapy in Acute Myeloid Leukemia Using 5hmC as a Blood-Based Minimal Residual Disease Marker
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Methodist Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO00038056 (HMCC-HM24-001)
Record Dates: First submitted 2025-06-20; First posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-06

CONDITIONS: Acute Myeloid Leukemia (AML); Acute Myeloid Leukaemia (AML)
Keywords: AML; Leukemia; Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia | interventions — venetoclax; Decitabine; Azacitidine; Cytarabine; Anthracyclines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- HMA- Based Treatment Arm (Active Comparator): Azacitidine or Decitabine with or without Venetoclax (HMA-based treatment):
  * Venetoclax is a BCL-2 inhibitor FDA Approved for the treatment of newly-diagnosed acute myeloid leukemia (AML) in adults who are age 75 years or older, or who have comorbidities that preclude use of intensive induction chemotherapy, in combination with azacitidine, decitabine or low-dose cytarabine in.
  * Decitabine is a nucleoside metabolic inhibitor that is administered as an intravenous infusion over a 1-3 hours.
  * Azacitidine can be given as a sub-cutaneous injection or intravenously. In AML, the most common adverse reactions (≥30%) in combination with azacitidine or decitabine or low-dose cytarabine were nausea, diarrhea, thrombocytopenia, constipation, neutropenia, febrile neutropenia, fatigue, vomiting, peripheral edema, pyrexia, pneumonia, dyspnea, hemorrhage, anemia, rash, abdominal pain, sepsis, back pain, myalgia, dizziness, cough, oropharyngeal pain, and hypotension.
  Interventions: Diagnostic Test: 5hmC Biomarker; Drug: Venetoclax; Drug: Decitabine 20 mg/m²/day for 5 days; Drug: Azacitidine (AZA)
- Intensive Chemotherapy Arm (Active Comparator): Cytarabine with Anthracycline (standard intensive induction therapy):
  * Cytarabine is FDA approved chemotherapy (pyrimidine analog) infusion that is frequently used with other drug such as anthracycline to treat acute myeloid leukemia, acute lymphoblastic leukemia. Common side effects include low counts, immune suppression, nausea, neutropenic fever.
  * Anthracyclines are chemotherapy infusions which topoisomerase II inhibition. Other than having side effects similar to cytarabine, it may cause weakening of heart pumping function few years later. Both of these medications may cause a temporary loss of hair in some people. After treatment with cytarabine has ended, normal hair growth should return.
  Interventions: Diagnostic Test: 5hmC Biomarker; Drug: Cytarabine (Ara-C); Drug: Anthracycline

INTERVENTIONS:
Diagnostic Test: 5hmC Biomarker — The 5hmC marker will be used to determine treatment modality post-induction therapy. After Week 4 of standard-of-care therapy (either HMA-based treatment or intensive induction chemotherapy), 5hmC biomarker testing will be performed. If MRD is positive, patients will continue the same standard-of-care treatment or crossover to the other arm of the study. If MRD is negative, patients will proceed with consolidation (either HSCT or continue on same treatment). For patients receiving HMA-based treatment, blood samples will be collected ± 5 days before and after 4 and 12 weeks of therapy. For patients receiving intensive chemotherapy blood samples will be collected ± 5 days before and after 4 and 12 weeks of therapy.
Drug: Venetoclax — Venetoclax is a BCL-2 inhibitor FDA Approved for the treatment of newly-diagnosed acute myeloid leukemia (AML) in adults who are age 75 years or older, or who have comorbidities that preclude use of intensive induction chemotherapy, in combination with azacitidine, decitabine or low-dose cytarabine.
  Arms: HMA- Based Treatment Arm
Drug: Decitabine 20 mg/m²/day for 5 days — Decitabine is a nucleoside metabolic inhibitor that is administered as an intravenous infusion over a 1-3 hours.
  Arms: HMA- Based Treatment Arm
Drug: Azacitidine (AZA) — Azacitidine can be given as a sub-cutaneous injection or intravenously.
  Arms: HMA- Based Treatment Arm
Drug: Cytarabine (Ara-C) — Cytarabine is FDA approved chemotherapy (pyrimidine analog) infusion that is frequently used with other drug such as anthracycline to treat acute myeloid leukemia, acute lymphoblastic leukemia. Common side effects include low counts, immune suppression, nausea, neutropenic fever.
  Arms: Intensive Chemotherapy Arm
Drug: Anthracycline — Anthracyclines are chemotherapy infusions which topoisomerase II inhibition. Other than having side effects similar to cytarabine, it may cause weakening of heart pumping function few years later. Both of these medications may cause a temporary loss of hair in some people. After treatment with cytarabine has ended, normal hair growth should return.
  Arms: Intensive Chemotherapy Arm

SUMMARY:
This is a therapeutic intervention trial evaluating the clinical utility of a novel blood-based epigenetic biomarker-genome-wide 5-hydroxymethylcytosine (5hmC) in cell-free DNA (cfDNA)-for assessing measurable residual disease (MRD) in patients with newly diagnosed acute myeloid leukemia (AML). The study compares the efficacy of hypomethylating agent (HMA)-based therapy versus intensive induction chemotherapy, using the 5hmC biomarker to guide post-induction treatment decisions. Approximately 112 adult patients will be enrolled and assigned to treatment arms based on a stratified sampling scheme. Blood samples will be collected at defined intervals to assess MRD status. Primary endpoints include minimal residual disease (MRD) negativity rate, duration of remission, event-free survival (EFS), and overall survival (OS).

DETAILED DESCRIPTION:
This is a therapeutic intervention trial evaluating the efficacy of a novel, blood epigenetic marker [genome-wide 5 hydroxymethylcytosine (5hmC) of cell free DNA (cfDNA)] for assessing measurable residual disease (MRD) in patients with acute myeloid leukemia (AML). Using the highly sensitive cfDNA 5hmC method, the trial will evaluate clinical efficacy of induction therapy and minimal residual disease (MRD) guided therapy in AML patients. Female or male patients aged 18 years, or older, with newly diagnosed de novo AML who will receive induction therapy with either hypomethylating agent (HMA) -based treatment or intensive chemotherapy will be eligible to participate in the trial. Patients will be assigned to one of the two treatment options based on a stratified sampling scheme. Approximately, 112 patients will be enrolled in the study. Informed consent will be obtained from all patients prior to participation.

The efficacy of HMA-based treatment versus intensive induction chemotherapy will be evaluated using the cfDNA 5hmC method in AML patients. The 5hmC marker will be used to determine treatment modality post-induction therapy. After Week 4 of standard-of-care therapy (either HMA-based treatment or intensive induction chemotherapy), 5hmC biomarker testing will be performed. If MRD is positive, patients will continue the same standard-of-care treatment or crossover to the other arm of the study. If MRD is negative, patients will proceed with consolidation (either HSCT or continue on same treatment).

For patients receiving HMA-based treatment, blood samples will be collected ± 5 days before and after 4 and 12 weeks of therapy. For patients receiving intensive chemotherapy blood samples will be collected ± 5 days before and after 4 and 12 weeks of therapy. The primary endpoints will be assessment of cfDNA 5hmC-MRD negativity rate, duration of remission, event-free survival (EFS), and overall survival (OS) in the two treatment groups. EFS will be assessed from the time of treatment initiation to the first occurrence of disease progression (>5% blasts in blood or bone marrow) or death from any cause. All sample collections will be conducted in accordance with the patient's standard-of-care visits. Patient samples will be collected prospectively at Houston Methodist Hospital. At least 112 subjects will be enrolled.

The hypothesis is that the 5hmC method for MRD detection will be more sensitive in AML patients receiving HMA-based regimens compared with those receiving intensive induction chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. The patient (or legally acceptable representative if applicable) provides written informed consent for the trial. Spanish speaking patients will be included and translation services will be provided as needed.
2. Male or female, 18 years of age or older, on the day of informed consent signing.
3. Newly diagnosed de novo AML

5. Expected life expectancy of at least 6 months 6. Willing and able to comply with the protocol for the duration of the trial including undergoing treatment and scheduled visits and examinations. 7. Women with childbearing potential and men should practice at least one of the following methods of birth control throughout the study and for 6 for women and 3 months for men after the last dose of study therapy:

1. Total abstinence from sexual intercourse (periodic abstinence not acceptable);
2. Surgically sterile partner(s) including vasectomy, bilateral tubal ligation, bilateral oophorectomy, or hysterectomy;
3. Practicing 2 effective methods of contraception (at least 1 highly effective, method of contraception [See Appendix 4]). WOCBP should only be included after a confirmed negative serum pregnancy test.

Exclusion Criteria:

1. Currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 3 weeks of trial treatment administration.
2. The patient has serious and/or uncontrolled preexisting medical condition(s) that, in the judgment of the investigator, would preclude participation in this study
3. Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
4. Confirmed positive pregnancy test in WOCBP.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 112 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
5hmC Minimal Residual Disease Rates | From date of initial treatment until progression, unacceptable toxicity, treating physician's discretion, or patient withdraws, whichever comes first, assessed up to 30 months.
  cfDNA 5hmC-MRD negativity and positivity rates at the time of morphologic remission.
Duration of Remission (DoR) Based on 5hmC-MRD Status | From date of initial treatment until progression, unacceptable toxicity, treating physician's discretion, or patient withdraws, whichever comes first, assessed up to 30 months.
  Time from initial treatment to disease relapse or progression, stratified by 5-hydroxymethylcytosine minimal residual disease (5hmC-MRD) status (positive vs. negative). This measure evaluates the impact of 5hmC-MRD on the sustainability of remission.
Event-Free Survival (EFS) by 5hmC-MRD Status | From date of initial treatment until progression, unacceptable toxicity, treating physician's discretion, or patient withdraws, whichever comes first, assessed up to 30 months.
  Time from treatment initiation to the occurrence of any treatment failure event, including relapse, progression, or death from any cause, compared between patients with positive and negative 5hmC-MRD. This outcome assesses the prognostic value of 5hmC-MRD in predicting treatment durability.
Overall Survival (OS) in Relation to 5hmC-MRD | From date of initial treatment until progression, unacceptable toxicity, treating physician's discretion, or patient withdraws, whichever comes first, assessed up to 30 months.
  Time from diagnosis or treatment start to death from any cause, analyzed by 5hmC-MRD status. This outcome measure determines whether 5hmC-MRD positivity is associated with reduced overall survival.

SECONDARY OUTCOMES:
MRD Positivity Rate Across Detection Methods | From date of initial treatment until progression, unacceptable toxicity, treating physician's discretion, or patient withdraws, whichever comes first, assessed up to 30 months.
  Proportion of patients identified as MRD-positive following induction therapy using 5hmC, multiparameter flow cytometry (MFC), RT-PCR, and next-generation sequencing (NGS). This outcome compares the sensitivity and concordance of MRD detection methods.
Duration of Remission (DoR) in MRD-Positive and MRD-Negative Patients by Method | From date of initial treatment until progression, unacceptable toxicity, treating physician's discretion, or patient withdraws, whichever comes first, assessed up to 30 months.
  Time from initial treatment to relapse or progression, stratified by MRD status (positive vs. negative) as determined by 5hmC, MFC, RT-PCR, and NGS. This outcome evaluates the prognostic value of each method in predicting remission durability.
Event-Free Survival by MRD Detection Method | From date of initial treatment until progression, unacceptable toxicity, treating physician's discretion, or patient withdraws, whichever comes first, assessed up to 30 months.
  Event-free survival (EFS) measured from treatment initiation, stratified by MRD status as determined by each method (5hmC, MFC, RT-PCR, NGS). This outcome assesses the predictive utility of each MRD method for long-term clinical outcomes.
Overall Survival by MRD Detection Method | From date of initial treatment until progression, unacceptable toxicity, treating physician's discretion, or patient withdraws, whichever comes first, assessed up to 30 months.
  Overall survival (OS) measured from treatment initiation, stratified by MRD status as determined by each method (5hmC, MFC, RT-PCR, NGS). This outcome assesses the predictive utility of each MRD method for long-term clinical outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Shilpan Shah, MD, Principal Investigator — Houston Methodist Neal Cancer Center
Locations (1):
- Houston Methodist Neal Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data sets regarding the correlation between minimal residual disease using the 5hmC biomarker and the type of standard of care treatment may be used by researchers at Houston Methodist and/or shared with other researchers, the government, and other institutions for use in future research.

REFERENCES:
- [Background] Krug U, Rollig C, Koschmieder A, Heinecke A, Sauerland MC, Schaich M, Thiede C, Kramer M, Braess J, Spiekermann K, Haferlach T, Haferlach C, Koschmieder S, Rohde C, Serve H, Wormann B, Hiddemann W, Ehninger G, Berdel WE, Buchner T, Muller-Tidow C; German Acute Myeloid Leukaemia Cooperative Group; Study Alliance Leukemia Investigators. Complete remission and early death after intensive chemotherapy in patients aged 60 years or older with acute myeloid leukaemia: a web-based application for prediction of outcomes. Lancet. 2010 Dec 11;376(9757):2000-8. doi: 10.1016/S0140-6736(10)62105-8. Epub 2010 Dec 3. PMID 21131036
- [Background] Appelbaum FR, Gundacker H, Head DR, Slovak ML, Willman CL, Godwin JE, Anderson JE, Petersdorf SH. Age and acute myeloid leukemia. Blood. 2006 May 1;107(9):3481-5. doi: 10.1182/blood-2005-09-3724. Epub 2006 Feb 2. PMID 16455952
- [Background] Camus V, Stamatoullas A, Mareschal S, Viailly PJ, Sarafan-Vasseur N, Bohers E, Dubois S, Picquenot JM, Ruminy P, Maingonnat C, Bertrand P, Cornic M, Tallon-Simon V, Becker S, Veresezan L, Frebourg T, Vera P, Bastard C, Tilly H, Jardin F. Detection and prognostic value of recurrent exportin 1 mutations in tumor and cell-free circulating DNA of patients with classical Hodgkin lymphoma. Haematologica. 2016 Sep;101(9):1094-101. doi: 10.3324/haematol.2016.145102. Epub 2016 Jun 13. PMID 27479820
- [Background] Armand P, Oki Y, Neuberg DS, Faham M, Cummings C, Klinger M, Weng L, Bhattar S, Lacasce AS, Jacobsen ED, Davids MS, Jacobson C, Fisher DC, Brown JR, Fowler NH, Alma Rodriguez M, Wallace MJ, Neelapu SS, Rodig S, Younes A, Freedman AS. Detection of circulating tumour DNA in patients with aggressive B-cell non-Hodgkin lymphoma. Br J Haematol. 2013 Oct;163(1):123-6. doi: 10.1111/bjh.12439. Epub 2013 Jun 25. No abstract available. PMID 23795711
- [Background] Cuccaro A, Bartolomei F, Cupelli E, Galli E, Giachelia M, Hohaus S. Prognostic factors in hodgkin lymphoma. Mediterr J Hematol Infect Dis. 2014 Jul 5;6(1):e2014053. doi: 10.4084/MJHID.2014.053. eCollection 2014. PMID 25045461
- [Background] Schwarz AK, Stanulla M, Cario G, Flohr T, Sutton R, Moricke A, Anker P, Stroun M, Welte K, Bartram CR, Schrappe M, Schrauder A. Quantification of free total plasma DNA and minimal residual disease detection in the plasma of children with acute lymphoblastic leukemia. Ann Hematol. 2009 Sep;88(9):897-905. doi: 10.1007/s00277-009-0698-6. Epub 2009 Jan 23. PMID 19165483
- [Background] Nakamura S, Yokoyama K, Shimizu E, Yusa N, Kondoh K, Ogawa M, Takei T, Kobayashi A, Ito M, Isobe M, Konuma T, Kato S, Kasajima R, Wada Y, Nagamura-Inoue T, Yamaguchi R, Takahashi S, Imoto S, Miyano S, Tojo A. Prognostic impact of circulating tumor DNA status post-allogeneic hematopoietic stem cell transplantation in AML and MDS. Blood. 2019 Jun 20;133(25):2682-2695. doi: 10.1182/blood-2018-10-880690. Epub 2019 Apr 1. PMID 30936070
- [Background] Bohers E, Viailly PJ, Dubois S, Bertrand P, Maingonnat C, Mareschal S, Ruminy P, Picquenot JM, Bastard C, Desmots F, Fest T, Leroy K, Tilly H, Jardin F. Somatic mutations of cell-free circulating DNA detected by next-generation sequencing reflect the genetic changes in both germinal center B-cell-like and activated B-cell-like diffuse large B-cell lymphomas at the time of diagnosis. Haematologica. 2015 Jul;100(7):e280-4. doi: 10.3324/haematol.2015.123612. Epub 2015 Mar 6. No abstract available. PMID 25749829
- [Background] Yeh P, Dickinson M, Ftouni S, Hunter T, Sinha D, Wong SQ, Agarwal R, Vedururu R, Doig K, Fong CY, Blombery P, Westerman D, Dawson MA, Dawson SJ. Molecular disease monitoring using circulating tumor DNA in myelodysplastic syndromes. Blood. 2017 Mar 23;129(12):1685-1690. doi: 10.1182/blood-2016-09-740308. Epub 2017 Jan 26. PMID 28126926
- [Background] Suzuki Y, Tomita A, Nakamura F, Iriyama C, Shirahata-Adachi M, Shimada K, Akashi A, Ishikawa Y, Kaneda N, Kiyoi H. Peripheral blood cell-free DNA is an alternative tumor DNA source reflecting disease status in myelodysplastic syndromes. Cancer Sci. 2016 Sep;107(9):1329-37. doi: 10.1111/cas.12994. Epub 2016 Aug 25. PMID 27323954
- [Background] Quan J, Gao YJ, Yang ZL, Chen H, Xian JR, Zhang SS, Zou Q, Zhang L. Quantitative detection of circulating nucleophosmin mutations DNA in the plasma of patients with acute myeloid leukemia. Int J Med Sci. 2015 Jan 1;12(1):17-22. doi: 10.7150/ijms.10144. eCollection 2015. PMID 25552914
- [Background] Albitar F, Ma W, Diep K, De Dios I, Agersborg S, Thangavelu M, Brodie S, Albitar M. Deep Sequencing of Cell-Free Peripheral Blood DNA as a Reliable Method for Confirming the Diagnosis of Myelodysplastic Syndrome. Genet Test Mol Biomarkers. 2016 Jul;20(7):341-5. doi: 10.1089/gtmb.2015.0278. Epub 2016 Jun 1. PMID 27248906
- [Background] Iriyama C, Tomita A, Hoshino H, Adachi-Shirahata M, Furukawa-Hibi Y, Yamada K, Kiyoi H, Naoe T. Using peripheral blood circulating DNAs to detect CpG global methylation status and genetic mutations in patients with myelodysplastic syndrome. Biochem Biophys Res Commun. 2012 Mar 23;419(4):662-9. doi: 10.1016/j.bbrc.2012.02.071. Epub 2012 Feb 20. PMID 22382018
- [Background] Vasioukhin V, Anker P, Maurice P, Lyautey J, Lederrey C, Stroun M. Point mutations of the N-ras gene in the blood plasma DNA of patients with myelodysplastic syndrome or acute myelogenous leukaemia. Br J Haematol. 1994 Apr;86(4):774-9. doi: 10.1111/j.1365-2141.1994.tb04828.x. PMID 7918071
- [Background] Buedts L, Vandenberghe P. Circulating cell-free DNA in hematological malignancies. Haematologica. 2016 Sep;101(9):997-9. doi: 10.3324/haematol.2015.131128. No abstract available. PMID 27582567
- [Background] Kubaczkova V, Vrabel D, Sedlarikova L, Besse L, Sevcikova S. Cell-free DNA - Minimally invasive marker of hematological malignancies. Eur J Haematol. 2017 Oct;99(4):291-299. doi: 10.1111/ejh.12925. Epub 2017 Aug 3. PMID 28692178
- [Background] Shao J, Shah S, Ganguly S, Zu Y, He C, Li Z. Classification of Acute Myeloid Leukemia by Cell-Free DNA 5-Hydroxymethylcytosine. Genes (Basel). 2023 May 28;14(6):1180. doi: 10.3390/genes14061180. PMID 37372359
- [Background] Shao J, Shah S, Ganguly S, Zu Y, He C, Li Z. Cell-free DNA 5-hydroxymethylcytosine is highly sensitive for MRD assessment in acute myeloid leukemia. Clin Epigenetics. 2023 Aug 24;15(1):134. doi: 10.1186/s13148-023-01547-0. PMID 37620919
- [Background] Shao J, Wang S, West-Szymanski D, Karpus J, Shah S, Ganguly S, Smith J, Zu Y, He C, Li Z. Cell-free DNA 5-hydroxymethylcytosine is an emerging marker of acute myeloid leukemia. Sci Rep. 2022 Jul 20;12(1):12410. doi: 10.1038/s41598-022-16685-3. PMID 35859008
- [Background] Shao J, Olsen RJ, Kasparian S, He C, Bernicker EH, Li Z. Cell-Free DNA 5-Hydroxymethylcytosine Signatures for Lung Cancer Prognosis. Cells. 2024 Feb 6;13(4):298. doi: 10.3390/cells13040298. PMID 38391911
- [Background] Xiao Z, Wu W, Wu C, Li M, Sun F, Zheng L, Liu G, Li X, Yun Z, Tang J, Yu Y, Luo S, Sun W, Feng X, Cheng Q, Tao X, Wu S, Tao J. 5-Hydroxymethylcytosine signature in circulating cell-free DNA as a potential diagnostic factor for early-stage colorectal cancer and precancerous adenoma. Mol Oncol. 2021 Jan;15(1):138-150. doi: 10.1002/1878-0261.12833. Epub 2020 Nov 14. PMID 33107199
- [Background] Guler GD, Ning Y, Ku CJ, Phillips T, McCarthy E, Ellison CK, Bergamaschi A, Collin F, Lloyd P, Scott A, Antoine M, Wang W, Chau K, Ashworth A, Quake SR, Levy S. Detection of early stage pancreatic cancer using 5-hydroxymethylcytosine signatures in circulating cell free DNA. Nat Commun. 2020 Oct 19;11(1):5270. doi: 10.1038/s41467-020-18965-w. PMID 33077732
- [Background] Tian X, Sun B, Chen C, Gao C, Zhang J, Lu X, Wang L, Li X, Xing Y, Liu R, Han X, Qi Z, Zhang X, He C, Han D, Yang YG, Kan Q. Circulating tumor DNA 5-hydroxymethylcytosine as a novel diagnostic biomarker for esophageal cancer. Cell Res. 2018 May;28(5):597-600. doi: 10.1038/s41422-018-0014-x. Epub 2018 Feb 21. No abstract available. PMID 29467383
- [Background] Cai J, Chen L, Zhang Z, Zhang X, Lu X, Liu W, Shi G, Ge Y, Gao P, Yang Y, Ke A, Xiao L, Dong R, Zhu Y, Yang X, Wang J, Zhu T, Yang D, Huang X, Sui C, Qiu S, Shen F, Sun H, Zhou W, Zhou J, Nie J, Zeng C, Stroup EK, Zhang X, Chiu BC, Lau WY, He C, Wang H, Zhang W, Fan J. Genome-wide mapping of 5-hydroxymethylcytosines in circulating cell-free DNA as a non-invasive approach for early detection of hepatocellular carcinoma. Gut. 2019 Dec;68(12):2195-2205. doi: 10.1136/gutjnl-2019-318882. Epub 2019 Jul 29. PMID 31358576
- [Background] Chiu BC, Zhang Z, You Q, Zeng C, Stepniak E, Bracci PM, Yu K, Venkataraman G, Smith SM, He C, Zhang W. Prognostic implications of 5-hydroxymethylcytosines from circulating cell-free DNA in diffuse large B-cell lymphoma. Blood Adv. 2019 Oct 8;3(19):2790-2799. doi: 10.1182/bloodadvances.2019000175. PMID 31570490
- [Background] Zhang J, Han X, Gao C, Xing Y, Qi Z, Liu R, Wang Y, Zhang X, Yang YG, Li X, Sun B, Tian X. 5-Hydroxymethylome in Circulating Cell-free DNA as A Potential Biomarker for Non-small-cell Lung Cancer. Genomics Proteomics Bioinformatics. 2018 Jun;16(3):187-199. doi: 10.1016/j.gpb.2018.06.002. Epub 2018 Jul 18. PMID 30010036
- [Background] Li W, Zhang X, Lu X, You L, Song Y, Luo Z, Zhang J, Nie J, Zheng W, Xu D, Wang Y, Dong Y, Yu S, Hong J, Shi J, Hao H, Luo F, Hua L, Wang P, Qian X, Yuan F, Wei L, Cui M, Zhang T, Liao Q, Dai M, Liu Z, Chen G, Meckel K, Adhikari S, Jia G, Bissonnette MB, Zhang X, Zhao Y, Zhang W, He C, Liu J. 5-Hydroxymethylcytosine signatures in circulating cell-free DNA as diagnostic biomarkers for human cancers. Cell Res. 2017 Oct;27(10):1243-1257. doi: 10.1038/cr.2017.121. Epub 2017 Sep 19. PMID 28925386
- [Background] Han D, Lu X, Shih AH, Nie J, You Q, Xu MM, Melnick AM, Levine RL, He C. A Highly Sensitive and Robust Method for Genome-wide 5hmC Profiling of Rare Cell Populations. Mol Cell. 2016 Aug 18;63(4):711-719. doi: 10.1016/j.molcel.2016.06.028. Epub 2016 Jul 28. PMID 27477909
- [Background] Lovkvist C, Dodd IB, Sneppen K, Haerter JO. DNA methylation in human epigenomes depends on local topology of CpG sites. Nucleic Acids Res. 2016 Jun 20;44(11):5123-32. doi: 10.1093/nar/gkw124. Epub 2016 Feb 29. PMID 26932361
- [Background] Liang G, Wang L, You Q, Cahill K, Chen C, Zhang W, Fulton N, Stock W, Odenike O, He C, Han D. Cellular Composition and 5hmC Signature Predict the Treatment Response of AML Patients to Azacitidine Combined with Chemotherapy. Adv Sci (Weinh). 2023 Aug;10(23):e2300445. doi: 10.1002/advs.202300445. Epub 2023 Jun 4. PMID 37271891
- [Background] Konstandin N, Bultmann S, Szwagierczak A, Dufour A, Ksienzyk B, Schneider F, Herold T, Mulaw M, Kakadia PM, Schneider S, Spiekermann K, Leonhardt H, Bohlander SK. Genomic 5-hydroxymethylcytosine levels correlate with TET2 mutations and a distinct global gene expression pattern in secondary acute myeloid leukemia. Leukemia. 2011 Oct;25(10):1649-52. doi: 10.1038/leu.2011.134. Epub 2011 May 31. No abstract available. PMID 21625234
- [Background] Chen S, Zhou Q, Liu T, Zhang W, Zeng XT, Guo Z. Prognostic value of downregulated 5-hydroxymethylcytosine expression in renal cell carcinoma: a 10 year follow-up retrospective study. J Cancer. 2020 Jan 1;11(5):1212-1222. doi: 10.7150/jca.38283. eCollection 2020. PMID 31956367
- [Background] Wang Z, Du M, Yuan Q, Guo Y, Hutchinson JN, Su L, Zheng Y, Wang J, Mucci LA, Lin X, Hou L, Christiani DC. Epigenomic analysis of 5-hydroxymethylcytosine (5hmC) reveals novel DNA methylation markers for lung cancers. Neoplasia. 2020 Mar;22(3):154-161. doi: 10.1016/j.neo.2020.01.001. Epub 2020 Feb 12. PMID 32062069
- [Background] Tucker DW, Getchell CR, McCarthy ET, Ohman AW, Sasamoto N, Xu S, Ko JY, Gupta M, Shafrir A, Medina JE, Lee JJ, MacDonald LA, Malik A, Hasselblatt KT, Li W, Zhang H, Kaplan SJ, Murphy GF, Hirsch MS, Liu JF, Matulonis UA, Terry KL, Lian CG, Dinulescu DM. Epigenetic Reprogramming Strategies to Reverse Global Loss of 5-Hydroxymethylcytosine, a Prognostic Factor for Poor Survival in High-grade Serous Ovarian Cancer. Clin Cancer Res. 2018 Mar 15;24(6):1389-1401. doi: 10.1158/1078-0432.CCR-17-1958. Epub 2017 Dec 20. PMID 29263182
- [Background] Bosio M, Salvaterra E, Datturi F, Morbini P, Zorzetto M, Inghilleri S, Tomaselli S, Mangiarotti P, Meloni F, Cerveri I, Stella GM. 5-hydroxymethylcytosine but not MTAP methylation status can stratify malignant pleural mesothelioma based on the lineage of origin. Multidiscip Respir Med. 2018 Aug 2;13:27. doi: 10.1186/s40248-018-0137-4. eCollection 2018. PMID 30123503
- [Background] Tong M, Gao S, Qi W, Shi C, Qiu M, Yang F, Bai S, Li H, Wang Z, Sun Z, Wang L, Che Y. 5-Hydroxymethylcytosine as a potential epigenetic biomarker in papillary thyroid carcinoma. Oncol Lett. 2019 Sep;18(3):2304-2309. doi: 10.3892/ol.2019.10531. Epub 2019 Jun 27. PMID 31452729
- [Background] Applebaum MA, Barr EK, Karpus J, Nie J, Zhang Z, Armstrong AE, Uppal S, Sukhanova M, Zhang W, Chlenski A, Salwen HR, Wilkinson E, Dobratic M, Grossman R, Godley LA, Stranger BE, He C, Cohn SL. 5-Hydroxymethylcytosine Profiles Are Prognostic of Outcome in Neuroblastoma and Reveal Transcriptional Networks That Correlate With Tumor Phenotype. JCO Precis Oncol. 2019;3:PO.18.00402. doi: 10.1200/PO.18.00402. Epub 2019 May 16. PMID 31179414
- [Background] Liu J, Jiang J, Mo J, Liu D, Cao D, Wang H, He Y, Wang H. Global DNA 5-Hydroxymethylcytosine and 5-Formylcytosine Contents Are Decreased in the Early Stage of Hepatocellular Carcinoma. Hepatology. 2019 Jan;69(1):196-208. doi: 10.1002/hep.30146. Epub 2018 Dec 17. PMID 30070373
- [Background] Lemonnier F, Poullot E, Dupuy A, Couronne L, Martin N, Scourzic L, Fataccioli V, Bruneau J, Cairns RA, Mak TW, Bernard OA, de Leval L, Gaulard P. Loss of 5-hydroxymethylcytosine is a frequent event in peripheral T-cell lymphomas. Haematologica. 2018 Mar;103(3):e115-e118. doi: 10.3324/haematol.2017.167973. Epub 2017 Dec 14. No abstract available. PMID 29242297
- [Background] Qiu L, Liu F, Yi S, Li X, Liu X, Xiao C, Lian CG, Tu P, Wang Y. Loss of 5-Hydroxymethylcytosine Is an Epigenetic Biomarker in Cutaneous T-Cell Lymphoma. J Invest Dermatol. 2018 Nov;138(11):2388-2397. doi: 10.1016/j.jid.2018.05.007. Epub 2018 May 24. PMID 29803640
- [Background] Wernig-Zorc S, Yadav MP, Kopparapu PK, Bemark M, Kristjansdottir HL, Andersson PO, Kanduri C, Kanduri M. Global distribution of DNA hydroxymethylation and DNA methylation in chronic lymphocytic leukemia. Epigenetics Chromatin. 2019 Jan 7;12(1):4. doi: 10.1186/s13072-018-0252-7. PMID 30616658
- [Background] Liu X, Zhang G, Yi Y, Xiao L, Pei M, Liu S, Luo Y, Zhong H, Xu Y, Zheng W, Shen J. Decreased 5-hydroxymethylcytosine levels are associated with TET2 mutation and unfavorable overall survival in myelodysplastic syndromes. Leuk Lymphoma. 2013 Nov;54(11):2466-73. doi: 10.3109/10428194.2013.778408. Epub 2013 Mar 27. PMID 23432690
- [Background] Bowman RL, Levine RL. TET2 in Normal and Malignant Hematopoiesis. Cold Spring Harb Perspect Med. 2017 Aug 1;7(8):a026518. doi: 10.1101/cshperspect.a026518. PMID 28242787
- [Background] Ko M, Huang Y, Jankowska AM, Pape UJ, Tahiliani M, Bandukwala HS, An J, Lamperti ED, Koh KP, Ganetzky R, Liu XS, Aravind L, Agarwal S, Maciejewski JP, Rao A. Impaired hydroxylation of 5-methylcytosine in myeloid cancers with mutant TET2. Nature. 2010 Dec 9;468(7325):839-43. doi: 10.1038/nature09586. PMID 21057493
- [Background] Kroeze LI, Aslanyan MG, van Rooij A, Koorenhof-Scheele TN, Massop M, Carell T, Boezeman JB, Marie JP, Halkes CJ, de Witte T, Huls G, Suciu S, Wevers RA, van der Reijden BA, Jansen JH; EORTC Leukemia Group and GIMEMA. Characterization of acute myeloid leukemia based on levels of global hydroxymethylation. Blood. 2014 Aug 14;124(7):1110-8. doi: 10.1182/blood-2013-08-518514. Epub 2014 Jul 1. PMID 24986689
- [Background] Chen K, Zhang J, Guo Z, Ma Q, Xu Z, Zhou Y, Xu Z, Li Z, Liu Y, Ye X, Li X, Yuan B, Ke Y, He C, Zhou L, Liu J, Ci W. Loss of 5-hydroxymethylcytosine is linked to gene body hypermethylation in kidney cancer. Cell Res. 2016 Jan;26(1):103-18. doi: 10.1038/cr.2015.150. Epub 2015 Dec 18. PMID 26680004
- [Background] Xu T, Gao H. Hydroxymethylation and tumors: can 5-hydroxymethylation be used as a marker for tumor diagnosis and treatment? Hum Genomics. 2020 May 6;14(1):15. doi: 10.1186/s40246-020-00265-5. PMID 32375881
- [Background] Zeng C, Stroup EK, Zhang Z, Chiu BC, Zhang W. Towards precision medicine: advances in 5-hydroxymethylcytosine cancer biomarker discovery in liquid biopsy. Cancer Commun (Lond). 2019 Mar 29;39(1):12. doi: 10.1186/s40880-019-0356-x. PMID 30922396
- [Background] Vonk CM, Al Hinai ASA, Hanekamp D, Valk PJM. Molecular Minimal Residual Disease Detection in Acute Myeloid Leukemia. Cancers (Basel). 2021 Oct 29;13(21):5431. doi: 10.3390/cancers13215431. PMID 34771594
- [Background] Buldini B, Maurer-Granofszky M, Varotto E, Dworzak MN. Flow-Cytometric Monitoring of Minimal Residual Disease in Pediatric Patients With Acute Myeloid Leukemia: Recent Advances and Future Strategies. Front Pediatr. 2019 Oct 11;7:412. doi: 10.3389/fped.2019.00412. eCollection 2019. PMID 31681710
- [Background] Short NJ, Zhou S, Fu C, Berry DA, Walter RB, Freeman SD, Hourigan CS, Huang X, Nogueras Gonzalez G, Hwang H, Qi X, Kantarjian H, Ravandi F. Association of Measurable Residual Disease With Survival Outcomes in Patients With Acute Myeloid Leukemia: A Systematic Review and Meta-analysis. JAMA Oncol. 2020 Dec 1;6(12):1890-1899. doi: 10.1001/jamaoncol.2020.4600. PMID 33030517
- [Background] Dohner H, Estey E, Grimwade D, Amadori S, Appelbaum FR, Buchner T, Dombret H, Ebert BL, Fenaux P, Larson RA, Levine RL, Lo-Coco F, Naoe T, Niederwieser D, Ossenkoppele GJ, Sanz M, Sierra J, Tallman MS, Tien HF, Wei AH, Lowenberg B, Bloomfield CD. Diagnosis and management of AML in adults: 2017 ELN recommendations from an international expert panel. Blood. 2017 Jan 26;129(4):424-447. doi: 10.1182/blood-2016-08-733196. Epub 2016 Nov 28. PMID 27895058
- [Background] Dohner H, Wei AH, Appelbaum FR, Craddock C, DiNardo CD, Dombret H, Ebert BL, Fenaux P, Godley LA, Hasserjian RP, Larson RA, Levine RL, Miyazaki Y, Niederwieser D, Ossenkoppele G, Rollig C, Sierra J, Stein EM, Tallman MS, Tien HF, Wang J, Wierzbowska A, Lowenberg B. Diagnosis and management of AML in adults: 2022 recommendations from an international expert panel on behalf of the ELN. Blood. 2022 Sep 22;140(12):1345-1377. doi: 10.1182/blood.2022016867. PMID 35797463
- [Background] Heuser M, Freeman SD, Ossenkoppele GJ, Buccisano F, Hourigan CS, Ngai LL, Tettero JM, Bachas C, Baer C, Bene MC, Bucklein V, Czyz A, Denys B, Dillon R, Feuring-Buske M, Guzman ML, Haferlach T, Han L, Herzig JK, Jorgensen JL, Kern W, Konopleva MY, Lacombe F, Libura M, Majchrzak A, Maurillo L, Ofran Y, Philippe J, Plesa A, Preudhomme C, Ravandi F, Roumier C, Subklewe M, Thol F, van de Loosdrecht AA, van der Reijden BA, Venditti A, Wierzbowska A, Valk PJM, Wood BL, Walter RB, Thiede C, Dohner K, Roboz GJ, Cloos J. 2021 Update on MRD in acute myeloid leukemia: a consensus document from the European LeukemiaNet MRD Working Party. Blood. 2021 Dec 30;138(26):2753-2767. doi: 10.1182/blood.2021013626. PMID 34724563
- [Background] Voso MT, Ottone T, Lavorgna S, Venditti A, Maurillo L, Lo-Coco F, Buccisano F. MRD in AML: The Role of New Techniques. Front Oncol. 2019 Jul 23;9:655. doi: 10.3389/fonc.2019.00655. eCollection 2019. PMID 31396481
- [Background] Burnett A, Wetzler M, Lowenberg B. Therapeutic advances in acute myeloid leukemia. J Clin Oncol. 2011 Feb 10;29(5):487-94. doi: 10.1200/JCO.2010.30.1820. Epub 2011 Jan 10. PMID 21220605
- [Background] Bloomfield CD, Lawrence D, Byrd JC, Carroll A, Pettenati MJ, Tantravahi R, Patil SR, Davey FR, Berg DT, Schiffer CA, Arthur DC, Mayer RJ. Frequency of prolonged remission duration after high-dose cytarabine intensification in acute myeloid leukemia varies by cytogenetic subtype. Cancer Res. 1998 Sep 15;58(18):4173-9. PMID 9751631
- [Background] Lancet JE, Uy GL, Cortes JE, Newell LF, Lin TL, Ritchie EK, Stuart RK, Strickland SA, Hogge D, Solomon SR, Stone RM, Bixby DL, Kolitz JE, Schiller GJ, Wieduwilt MJ, Ryan DH, Hoering A, Banerjee K, Chiarella M, Louie AC, Medeiros BC. CPX-351 (cytarabine and daunorubicin) Liposome for Injection Versus Conventional Cytarabine Plus Daunorubicin in Older Patients With Newly Diagnosed Secondary Acute Myeloid Leukemia. J Clin Oncol. 2018 Sep 10;36(26):2684-2692. doi: 10.1200/JCO.2017.77.6112. Epub 2018 Jul 19. PMID 30024784
- [Background] Pautas C, Merabet F, Thomas X, Raffoux E, Gardin C, Corm S, Bourhis JH, Reman O, Turlure P, Contentin N, de Revel T, Rousselot P, Preudhomme C, Bordessoule D, Fenaux P, Terre C, Michallet M, Dombret H, Chevret S, Castaigne S. Randomized study of intensified anthracycline doses for induction and recombinant interleukin-2 for maintenance in patients with acute myeloid leukemia age 50 to 70 years: results of the ALFA-9801 study. J Clin Oncol. 2010 Feb 10;28(5):808-14. doi: 10.1200/JCO.2009.23.2652. Epub 2010 Jan 4. PMID 20048183
- [Background] Fernandez HF, Sun Z, Yao X, Litzow MR, Luger SM, Paietta EM, Racevskis J, Dewald GW, Ketterling RP, Bennett JM, Rowe JM, Lazarus HM, Tallman MS. Anthracycline dose intensification in acute myeloid leukemia. N Engl J Med. 2009 Sep 24;361(13):1249-59. doi: 10.1056/NEJMoa0904544. PMID 19776406
- [Background] Cancer Genome Atlas Research Network; Ley TJ, Miller C, Ding L, Raphael BJ, Mungall AJ, Robertson A, Hoadley K, Triche TJ Jr, Laird PW, Baty JD, Fulton LL, Fulton R, Heath SE, Kalicki-Veizer J, Kandoth C, Klco JM, Koboldt DC, Kanchi KL, Kulkarni S, Lamprecht TL, Larson DE, Lin L, Lu C, McLellan MD, McMichael JF, Payton J, Schmidt H, Spencer DH, Tomasson MH, Wallis JW, Wartman LD, Watson MA, Welch J, Wendl MC, Ally A, Balasundaram M, Birol I, Butterfield Y, Chiu R, Chu A, Chuah E, Chun HJ, Corbett R, Dhalla N, Guin R, He A, Hirst C, Hirst M, Holt RA, Jones S, Karsan A, Lee D, Li HI, Marra MA, Mayo M, Moore RA, Mungall K, Parker J, Pleasance E, Plettner P, Schein J, Stoll D, Swanson L, Tam A, Thiessen N, Varhol R, Wye N, Zhao Y, Gabriel S, Getz G, Sougnez C, Zou L, Leiserson MD, Vandin F, Wu HT, Applebaum F, Baylin SB, Akbani R, Broom BM, Chen K, Motter TC, Nguyen K, Weinstein JN, Zhang N, Ferguson ML, Adams C, Black A, Bowen J, Gastier-Foster J, Grossman T, Lichtenberg T, Wise L, Davidsen T, Demchok JA, Shaw KR, Sheth M, Sofia HJ, Yang L, Downing JR, Eley G. Genomic and epigenomic landscapes of adult de novo acute myeloid leukemia. N Engl J Med. 2013 May 30;368(22):2059-74. doi: 10.1056/NEJMoa1301689. Epub 2013 May 1. PMID 23634996
- [Background] Yang X, Wong MPM, Ng RK. Aberrant DNA Methylation in Acute Myeloid Leukemia and Its Clinical Implications. Int J Mol Sci. 2019 Sep 16;20(18):4576. doi: 10.3390/ijms20184576. PMID 31527484
- [Background] Zjablovskaja P, Florian MC. Acute Myeloid Leukemia: Aging and Epigenetics. Cancers (Basel). 2019 Dec 31;12(1):103. doi: 10.3390/cancers12010103. PMID 31906064